CLINICAL TRIAL: NCT04705961
Title: Bile Leakage Test in Emergency Hydatid Liver Cyst Surgery Case Report
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Uylas, Principal Investigator, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: 10012021
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Surgery--Complications
Keywords: Hydatidosis; complications; intra-biliary rupture; biliary duct; echinococcus; echinococcosis
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In liver cyst hydatid surgery, presence of cysto-biliary communication (CBC) is important for the prevention of postoperative morbidity. If cysto-biliary connections are not obvious, diagnosis is not easy. Intraoperative bile leakage test has been shown to reduce postoperative biliary complications by revealing occult CBCs. However, bile leakage testing in emergency conditions such as hydatid cyst perforation has not been experienced so far.

DETAILED DESCRIPTION:
In liver cyst hydatid surgery, presence of cysto-biliary communication (CBC) is important for the prevention of postoperative morbidity. If cysto-biliary connections are not obvious, diagnosis is not easy. Intraoperative bile leakage test has been shown to reduce postoperative biliary complications by revealing occult CBCs. However, bile leakage testing in emergency conditions such as hydatid cyst perforation has not been experienced so far.

Here, a bile leakage test performed in a 23-year-old male patient undergoing emergency surgery due to the perforation of the hydatid liver cyst was presented. Following the treatment of perforated hydatid liver cyst and biliary peritonitis, a bile leakage test was performed. The common bile duct was cannulated with a 22 Gauge catheter, normal saline and parenteral lipid solution were given to demonstrate the CBCs, and leakage areas were suture ligated. The patient was discharged postoperatively without any problem.

The investigators recommend detection and treatment of the CBCs even in emergency hydatid liver cyst surgery for prevention of postoperative biliary complications.

ELIGIBILITY:
Inclusion Criteria:

* this study is a case report

Exclusion Criteria:

* this study is a case report

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: this study is a case report
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
recurrent hydatid cyst | 2 or 3 month
  presence of recurrent hydatid cyst

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No